CLINICAL TRIAL: NCT04048603
Title: A 7-year Prospective Study of Idiopathic REM Sleep Behavior Disorder Cohort in Chinese Population: Determining the Optimal Characteristics of Biomarkers to Predict Neurodegenerative Diseases
Brief Title: Search for Biomarkers of Neurodegenerative Diseases in Idiopathic REM Sleep Behavior Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Zhang Jihui, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: 2018.641
Record Dates: First submitted 2019-03-22; First posted 2019-08-07 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: REM Sleep Behavior Disorder; Neurodegeneration
Keywords: REM sleep behavior disorder; Neurodegeneration; α-synucleinopathy; Prodromal markers
MeSH Terms: conditions — REM Sleep Behavior Disorder; Nerve Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Thyroid Function Tests(TFT), Vitamin B12, Folate, Complete Blood Count(CBC), Fasting Glucose, Liver Function Tests(LFT), Renal Function Tests(RFT), C-reactive protein(CRP), Fasting lipid, Iron profile, Phosphate, Calcium, Neurosteroid, Genetic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- idiopathic REM sleep behavior disorder: Subjects with the diagnosis of idiopathic REM sleep behavior disorder
- Controls without iRBD: Healthy controls without the diagnosis of idiopathic REM sleep behavior disorder

SUMMARY:
This study is a prospective study with a mean of 7-year follow-up interval, aims to monitor the progression of α-synucleinopathy neurodegeneration by the evolution of prodromal markers and development of clinical disorders in patients with idiopathic REM Sleep Behavior Disorder (iRBD) and healthy controls.

DETAILED DESCRIPTION:
REM sleep behavior disorder (RBD) is a parasomnia characterized by dream enactment behaviors and REM sleep without muscle atonia (excessive EMG activity) during REM sleep.Increasing studies revealed that iRBD eventually converts to α-synucleinopathy, such as Parkinson's disease (PD), dementia with Lewy Bodies (DLB), and multiple system atrophy (MSA). Recent studies reported that over 80% of patients with iRBD eventually developed neurodegeneration at a mean interval of 14 years after iRBD onset or diagnosed. Thus, iRBD is regarded as a precursor of α-synucleinopathies. In addition to iRBD, a large series of other non-motor symptoms also present before the emergence of typical motor symptoms of PD, including autonomic dysfunction, olfactory loss, color vision impairment, neurocognitive impairment,neuroimaging of dopamine dysfunction, daytime sleepiness, and psychiatric disorders. In recent years, several longitudinal studies have found that patients with iRBD with a higher rate of these markers may have a faster progression of neurodegeneration. On the other hand, a variety of external risk factors of PD including environmental toxic exposure, lifestyle factors, and some medications have long been recognized, which affect numerous fundamental cellular processes by interaction with genetic predisposition.

However, several knowledge gaps still need further studies to uncover. First, few studies have explored the predictive value of dynamic change of biomarkers in prodromal stage of PD. Second, few previous prospective studies also employed a control group to compare the change of these prodromal markers between patients and healthy controls over time. Third, as some of previous studies employed a retrospective study design, potential recall bias may contaminate the results. Moreover, the sample sizes of most previous studies investigating biomarkers were relative small (n < 80) and follow-up durations in most study are relatively short, which may have limited the statistical power to detect the risk factors with mild to moderate effect size. Finally, as previous reported longitudinal studies of iRBD mainly focused on Caucasian or other ethnic groups, there is only limited data about neurodegenerative biomarkers in Chinese iRBD. In conclusion, prospective longitudinal studies with larger sample size, regular follow-up, and relative long follow-up duration are needed to better map the progression of neurodegeneration.

ELIGIBILITY:
Inclusion Criteria:

for iRBD at baseline:

1. Fulfilling the diagnostic criteria for iRBD. As patients with iRBD were recruited during a long period, the diagnosis of RBD was based on ICSD and ICSD-2 (before 2014), and ICSD-3 (2014 and thereafter) criteria. The diagnosis for all patients were confirmed by video-PSG. In summary, patient diagnosed with RBD should present excessive EMG activity during REM sleep on video-PSG assessment and report a history of repeated dream enactment behaviors;
2. Having neurocognitive test and neurological examination since 2008;
3. Free of neurodegenerative diseases at the last visit.

for controls without iRBD at baseline:

1. Age- and sex- matched with patients with iRBD;
2. Free of narcolepsy and other neurological diseases;
3. Without any RBD features as confirmed by both clinical history and video-PSG;
4. Without neurodegenerative diseases;
5. Having neurocognitive test and neurological examination at baseline.

Exclusion Criteria:

1. Patients with narcolepsy;
2. Patients with known neurodegenerative diseases;
3. Pseudo-RBD (e.g., RBD symptoms were eliminated after severe obstructive sleep apnea had treated with continuous positive airway pressure therapy.);
4. Early-onset RBD (e.g., before the age of 50 years old) which might have a different pathogenesis from iRBD.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants in this proposed study will be recruited from our on-going cohort of RBD and control
Sampling Method: Non-Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
The overall conversion rate of iRBD to neurodegenerative diseases | Changes from baseline to 7 year follow up
  The overall conversion rate of iRBD to neurodegenerative diseases. The diagnoses of neurodegenerative diseases will be ascertained by neurologists according to the standard diagnostic criteria.

SECONDARY OUTCOMES:
Changes of the likelihood ratio of probability of prodromal Parkinson's disease in each individual | Baseline and 7 year
  The dynamic changes of the likelihood ratio of probability of prodromal Parkinson's disease in the patients with iRBD and healthy controls will be calculated based on the Movement Disorder Society (MDS) research criteria for prodromal Parkinson's disease.
Conversion rate of iRBD to neurodegenerative diseases in patients with high and low likelihood ratio of probability of prodromal Parkinson's disease in each individual | Changes from baseline to 7 year follow up
  Conversion rate of iRBD to neurodegenerative diseases in patients with high and low likelihood ratio of probability at baseline, the level of likelihood ratio was defined based on the Movement Disorder Society (MDS) research criteria for prodromal Parkinson's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Zhang, PhD, Principal Investigator — Chinese University of Hong Kong; Yun Kwok Wing, MBChB, Study Director — Chinese University of Hong Kong; Yaping Liu, PhD, Study Director — Chinese University of Hong Kong; Siu Ping Lam, MBChB, Study Director — Chinese University of Hong Kong; Shirley Xin Li, PhD, Study Director — The University of Hong Kong; Vincent Chung Tong Mok, MBChB, Study Director — Chinese University of Hong Kong
Locations (1):
- Department of psychiatry, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Researcher in other sleep centers are also conducting similar study, there may be a plan for further collaboration on sharing the database